CLINICAL TRIAL: NCT04385589
Title: Safety and Efficacy of Adding Dapagliflozin and Furosemide in Diabetic Patients (Type 2) With Decompensated Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: Dapagliflozin in Diabetic Patients (Type 2) With Decompensated Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelfatah, principal investigator, Assiut University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 3241
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Insulin

STUDY DESIGN:
Intervention Model Description: The study will include 100 diabetic patients type 2 patients who will be admitted to care unit with decompensated heart failure.50 patient will receive Dapagliflozin plus insulin (if needed) and Diuretics plus conventional heart failure measures ,the other group will receive insulin for control of blood sugar plus diuretics and anti-failure measures.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Active Comparator): 50 patients will receive Dapagliflozin plus insulin (if needed) and Diuretics plus conventional heart failure measures.
  Interventions: Drug: Dapagliflozin; Drug: insulin
- Placebo group (Placebo Comparator): 50 patients will receive insulin for control of blood sugar plus diuretics and anti-failure measures.
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: Dapagliflozin — Patient will receive oral Dapagliflozin then monitoring of its efficacy on heart failure symptoms and outcome.
  Other Names: SGLT-2 inhibitors
  Arms: Dapagliflozin group
Drug: insulin — insulin

SUMMARY:
We hypothesize that Dapagliflozin could improve the diuretic response in diabetic patients with acute decompensated heart failure owing to its diuretic effect in addition to improvement of blood glucose level without remarkable effect on kidney function or electrolytes.

DETAILED DESCRIPTION:
The study will include 100 diabetic patients type 2 patients who will be admitted to care unit with decompensated heart failure.50 patient will receive Dapagliflozin plus insulin (if needed) and Diuretics plus conventional heart failure measures ,the other group will receive insulin for control of blood sugar plus diuretics and anti-failure measures.

Inclusion Criteria:

Diabetic patient type 2 with history of chronic heart failure(HFrEF) ,there is no specified inclusion criterion with respect to heart failure etiology and/or ejection fraction.

Age more than 18 years Admission for acute decompensated heart failure The patient already on an oral loop diuretic for at least 1 month before admission, at a dose between 40 mg and 80 mg daily in the case of furosemide and an equivalent dose in the case of a different loop diuretic (20 mg of Torsemide will be considered to be equivalent to 40 mg of furosemide.

Exclusion Criteria:

1. Other etiologies of fluid overload different from heart failure.
2. Hyponatremia: Sodium level below 125mmol/l
3. Unstable patients: acute coronary syndrome, cardiogenic shock .
4. Patients requiring inotropic agents or renal dialysis.
5. Pregnancy or breastfeeding period.
6. sever hepatic disease
7. GFR (Glomerular Filtration Rate) is less than 45 mL/min/1.73 m² .
8. Patient with diabetic ketoacidosis or non ketotic hyperosmolar. Treatment arm.

The patients will receive:

Loop diuretics. Diuretics should be administered at doses sufficient to achieve optimal volume status and relieve congestion without inducing an excessively rapid reduction in intravascular volume.

furosemide will be given I.V either by continuous infusion or blouses Antifailure treatment: (Angiotensin converting enzyme inhibitors or Angiotensin II Receptor Blockers, Beta Blockers,Mineralocorticoid Receptor Antagonists, Ivabradine, or others will be individualized according to the patient condition.

Dapagliflozin:

will be given in a dose of 10mg once daily ( GFR is more than 45 mL/min/1.73 m²) .

In Mild or moderate hepatic disease: No dosage adjustment required In Severe hepatic disease: will not be used.

Insulin. Insulin therapy should be initiated if blood glucose levels is ≥180 mg/dL (10.0 mmol/L) after initiation of Dapagliflozin treatment. Once insulin therapy is started, a target glucose range of 140-180 mg/dL (7.8-10.0 mmol/L) is recommended The use of subcutaneous rapid- or short-acting insulin before meals or every 4-6 h will be given to correct hyperglycemia according to sliding scale chart.

Control arm.

The patients will be given Loop diuretics. Anti-failure treatment. Insulin.

All the patients will undergo:

1. Complete echo assessment.
2. ECG on admission and daily.
3. Monitoring:24 hours ECG ,Oxygen saturation and blood pressure monitoring. Complete blood count ,blood urea,serum creatinine,blood sugar,electrolytes ,liver function will be measured on admission
4. Blood sugar ,urea,creatinine,Na, K will be measured daily along the whole days of admission.

Follow up parameters

Diuresis :24-hour diuresis will be quantified every 24 hours (during hospitalization) from the 1st day until last day of admission.

diuretic response will be measured by weight loss and net fluid loss per mg . Changes in body weight measurements: the mean of weight lost every 24 hours and the total weight lost from baseline to the last day of hospitalization Renal function will be determined every 24 hours (during hospitalization) from the date of admission until the date of discharge.

Renal function is assessed with the serum creatinine level. Worsening renal function is defined as an increase in the serum creatinine level of more than 0.3 mg/dl at any time during hospitalization Electrolyte levels (sodium and potassium) will be determined every 24 hours (during hospitalization) from the date of admission until the date of discharge.

Electrolyte levels are assessed with the serum sodium and potassium levels. Patient-reported dyspnea : Patient-reported dyspnea is assessed every 24 hours (during hospitalization) from the date of admission until the date of discharge.

Patient-reported dyspnea will be assessed with the use five point Linker scale.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient type 2 with history of chronic heart failure(HFrEF) ,there is no prespecified inclusion criterion with respect to heart failure etiology and/or ejection fraction.

Exclusion Criteria:

1. Other etiologies of fluid overload different from heart failure.
2. Hyponatremia: Sodium level below 125mmol/l
3. Unstable patients: acute coronary syndrome, cardiogenic shock .
4. Patients requiring inotropic agents or renal dialysis.
5. Pregnancy or breastfeeding period.
6. sever hepatic disease
7. GFR is less than 45 mL/min/1.73 m² .
8. Patient with diabetic ketoacidosis or non ketotic hyperosmolar.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in body weight measurement (Diuresis effect.) | Days of admission (3-5 days)
  Diuretic response will be measured by weight loss
Diuresis effect. | Days of admission (3-5 days)
  Diuretic response will be measured by net fluid loss per mg .

SECONDARY OUTCOMES:
Renal function | Days of admission (3-5 days)
  Renal function is assessed with the serum creatinine level. Worsening renal function is defined as an increase in the serum creatinine level of more than 0.3 mg/dl at any time during hospitalization
Patient-reported dyspnea will be assessed with the use five point Linker scale | Days of admission (3-5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Ibrahem, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohara K, Masuda T, Morinari M, Okada M, Miki A, Nakagawa S, Murakami T, Oka K, Asakura M, Miyazawa Y, Maeshima A, Akimoto T, Saito O, Nagata D. The extracellular volume status predicts body fluid response to SGLT2 inhibitor dapagliflozin in diabetic kidney disease. Diabetol Metab Syndr. 2020 May 1;12:37. doi: 10.1186/s13098-020-00545-z. eCollection 2020. PMID 32377235
- [Background] Elsisi GH, Anwar MM, Khattab M, Elebrashy I, Wafa A, Elhadad H, Awad M, Carapinha JL. Budget impact analysis for dapagliflozin in type 2 diabetes in Egypt. J Med Econ. 2020 Aug;23(8):908-914. doi: 10.1080/13696998.2020.1764571. Epub 2020 May 28. PMID 32364032
- [Background] Linden K, Mailey J, Kearney A, Menown IBA. Advances in Clinical Cardiology 2019: A Summary of Key Clinical Trials. Adv Ther. 2020 Jun;37(6):2620-2645. doi: 10.1007/s12325-020-01355-5. Epub 2020 May 2. PMID 32361851
- [Background] Cappetta D, De Angelis A, Ciuffreda LP, Coppini R, Cozzolino A, Micciche A, Dell'Aversana C, D'Amario D, Cianflone E, Scavone C, Santini L, Palandri C, Naviglio S, Crea F, Rota M, Altucci L, Rossi F, Capuano A, Urbanek K, Berrino L. Amelioration of diastolic dysfunction by dapagliflozin in a non-diabetic model involves coronary endothelium. Pharmacol Res. 2020 Jul;157:104781. doi: 10.1016/j.phrs.2020.104781. Epub 2020 Apr 28. PMID 32360273
- [Derived] Kasem SM, Saied GM, Hegazy ANM, Abdelsabour M. Impact of Acute Insulin Resistance on Myocardial Blush in Non-Diabetic Patients Undergoing Primary Percutaneous Coronary Intervention. Front Cardiovasc Med. 2021 May 10;8:647366. doi: 10.3389/fcvm.2021.647366. eCollection 2021. PMID 34041280
- [Derived] Ibrahim A, Ghaleb R, Mansour H, Hanafy A, Mahmoud NM, Abdelfatah Elsharef M, Kamal Salama M, Elsaughier SM, Abdel-Wahid L, Embarek Mohamed M, Ibrahim AK, Abdel-Galeel A. Safety and Efficacy of Adding Dapagliflozin to Furosemide in Type 2 Diabetic Patients With Decompensated Heart Failure and Reduced Ejection Fraction. Front Cardiovasc Med. 2020 Dec 7;7:602251. doi: 10.3389/fcvm.2020.602251. eCollection 2020. PMID 33426003